CLINICAL TRIAL: NCT01039662
Title: Effects of the Combination of L-Arabinose and Indigestible Dextrin on Glycemic Index: a Double-Blind, Crossover Trial
Brief Title: Reduction of the Dietary Glycemic Index (GI) by L-Arabinose and Indigestible Dextrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Unitika Ltd. (Industry)
Responsible Party: Fumiko Higashikawa, Associate professor, Hiroshima University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: eki-199
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
MeSH Terms: interventions — Arabinose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oolong tea containing L-arabinose and indigestible dextrin (Experimental)
  Interventions: Dietary Supplement: L-arabinose and indigestible dextrin
- Oolong tea (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-arabinose and indigestible dextrin
  Arms: Oolong tea containing L-arabinose and indigestible dextrin
Dietary Supplement: Placebo
  Arms: Oolong tea

SUMMARY:
This study aims to investigate the effect of supplement containing L-arabinose and indigestible dextrin on dietary glycemic index.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as based on medical history and physical examination
* BMI is less or equal to 30 kg/m2
* Willing not to serve as blood donor during the study
* Informed consent signed

Exclusion Criteria:

* Impaired Glucose Tolerance
* Female subjects who are pregnant or nursing a child
* Participation in any clinical trial up to 90 days before Day 1 of this study
* Renal or hepatic dysfunction
* Heart disease
* Under medication

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose level | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hiroshima University, Hiroshima, Hiroshima, Japan